CLINICAL TRIAL: NCT00584025
Title: Keppra IV for the Treatment of Motor Fluctuations in Parkinson's Disease
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study withdrawn due to personnel limitations.
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Theresa Zesiewicz, MD, Professor of Neurology, University of South Florida
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 5
Record Dates: First submitted 2007-12-21; First posted 2008-01-02 (Estimated); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; dyskinesia; levetiracetam; keppra
MeSH Terms: conditions — Parkinson Disease; Dyskinesias | interventions — Levetiracetam

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Keppra IV
  Interventions: Drug: levetiracetam
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: levetiracetam — 100 - 500mg IV q 15 min
  Arms: 1
Drug: Placebo — Placebo equivalent of 100 - 500 mg levetiracetam IV q 15 min
  Arms: 2

SUMMARY:
The primary purpose of this study is to characterize the acute anti-dyskinetic properties of intravenous levetiracetam in Parkinson's disease patients who have been optimized on antiparkinsonian medication. The secondary objective is to study the effect of intravenous LEV on additional motor and cognitive symptoms of PD.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients with idiopathic PD according to the UK Parkinson's Disease Society Brain Bank Clinical Diagnosis Criteria.
2. Age 30 years to 80 years.
3. Dyskinesias with a minimum severity equal to a rating of 10 or higher on the AIMS rating scale at baseline.
4. Dyskinesias at least moderately disabling (historical information from item 33 of UPDRS).
5. Stable dose of antiparkinsonian medication 4 weeks prior to study entry.
6. Women of child-bearing potential must use a reliable method of contraception and must be willing to perform a pregnancy test paid for and provided by Dr. Zesiewicz and the USF Medical Clinic. There must be a negative result before entry into the study.

Exclusion Criteria:

1. Any illness that in the investigator's opinion preclude participation in this study. This includes patients with unstable disease and those PD patients who can not tolerate IV infusion.
2. Pregnant or lactating women. Pregnancy will not be allowed whether as a pre-existing condition or a positive result on the pregnancy test in the screening process. Lactation includes any woman wanting to participate who is currently breast-feeding.
3. Patients may not be dual enrolled to another research study requiring the patient to sign informed consent.
4. Dementia or other psychiatric illness that prevents the patient from giving informed consent (Mini Mental Status Exam score of less than 20).
5. Legal incapacity or limited legal capacity.
6. Presence of severe renal disease (BUN 50% greater than normal). Patients must have evidence from their PCP or Urologists of normal PSA and urodynamic tests within the last 12 months; patients with BUN 50% greater than normal (5 to 20 mg/ d L) or creatinine 50% greater than normal (0 .7 and 1.4 mg/ d L) will be excluded. Labs will be requested from PCP.
7. Concomitant or prior therapy with the following treatments: neuroleptics, metoclopramide, domperidone (in doses >60mg/day), azole antifungals (e.g. ketoonazole), etomidate, ciprofloxacin, fluvoxamine, cimetidine, fludrocortizone, encainide, flecainide, mexiletine, propafenone, guanoxane, maprotiline, antidepressants on doses higher than the maximum approved daily dose for outpatients, intermittent therapy with oral corticoids.
8. Patients who are not fluent in English.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-12; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Abnormal Involuntary Movements Scale (AIMS) | 15 minutes

SECONDARY OUTCOMES:
Rush Dyskinesia Rating Scale | 15 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Theresa A Zesiewicz, MD, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States